CLINICAL TRIAL: NCT00537420
Title: A 24-Week, Blinded, Randomized, Placebo-Controlled Dose-Ranging Trial of Nasal PYY3-36 for Weight Loss in Healthy Obese Patients
Brief Title: A Study of Nasal PYY3-36 and Placebo for Weight Loss in Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nastech Pharmaceutical Company, Inc. (Industry)
Responsible Party: Gordon Brandt, M.D. / President, Nastech Pharmaceutical Company, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C07-002
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2008-09-15 (Estimated); Status verified 2008-09

CONDITIONS: Obesity
Keywords: weight loss; dieting
MeSH Terms: conditions — Obesity; Weight Loss | interventions — peptide YY (3-36); sibutramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Placebo Comparator): Nasal Placebo
  Interventions: Drug: Nasal Placebo
- 2 (Placebo Comparator): Capsule Placebo
  Interventions: Drug: Placebo Capsule
- 3 (Experimental): Nasal PYY3-36 200 ug
  Interventions: Drug: PYY3-36
- 4 (Experimental): Nasal PYY3-36 400 ug
  Interventions: Drug: PYY3-36
- 5 (Experimental): Nasal PYY3-36 600 ug
  Interventions: Drug: PYY3-36
- 6 (Active Comparator): Sibutramine 10 mg
  Interventions: Drug: Sibutramine

INTERVENTIONS:
Drug: Nasal Placebo — Nasal placebo, three times a day, 30 minutes before a meal for 24 weeks.
  Arms: 1
Drug: Placebo Capsule — Placebo capsules will be taken once daily with or without food.
  Arms: 2
Drug: PYY3-36 — Nasal PYY3-36, three times a day, 30 minutes before a meal for 24 weeks.
  Arms: 3
Drug: PYY3-36 — Nasal PYY3-36 three times a day, 30 minutes before a meal for 24 weeks.
  Arms: 4
Drug: PYY3-36 — Nasal PYY3-36 three times a day, 30 minutes before a meal for 24 weeks.
  Arms: 5
Drug: Sibutramine — Sibutramine will be taken once daily with or without food
  Other Names: Meridia
  Arms: 6

SUMMARY:
The purpose of this study is to determine the effect of nasal PYY3-36 on weight loss post 24 weeks of treatment.

DETAILED DESCRIPTION:
This is a multi-center, Phase 2 double-blind, randomized, placebo-controlled trial in healthy obese patients. The primary objective of the study is to evaluate the effect of increasing nasal PYY3-36 dosing on weight loss post 24 weeks of treatment.

Secondary Objectives:

* To evaluate the safety of three nasal PYY3 36 dose groups compared to nasal placebo
* To compare the weight loss post 12 and 24 weeks of treatment for each of the three nasal PYY3 36 dose groups versus the nasal placebo group
* To compare the proportion of patients who lose at least 5% and 10% of the baseline body weight post 12 and 24 weeks of therapy for each of the three nasal PYY3 36 dose groups versus the nasal placebo group
* To compare the weight loss and proportion of patients who lose at least 5% of the baseline body weight post 12 and 24 weeks of treatment with sibutramine versus capsule placebo
* To compare the weight loss and proportion of patients who lose at least 5% of the baseline body weight post 12 and 24 weeks of treatment with nasal placebo versus capsule placebo
* To compare the weight loss and proportion of patients who lose at least 5% of the baseline body weight post 12 and 24 weeks of treatment with sibutramine versus the nasal PYY3 36 dose groups
* To evaluate the effect of 12 and 24 weeks of treatment with nasal PYY3 36 and sibutramine on fasting lipid profile, plasma glucose, insulin, blood pressure and pulse, waist circumference and BMI
* To evaluate the effect of 24 weeks of treatment with nasal PYY3 36 and sibutramine on HbA1c levels

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients 18 and 65 years, inclusive;
* BMI 30-43 kg/m2, inclusive;
* In good health, determined by medical history and physical examination, as well as normal 12-lead ECG and vital signs;
* Non-smoker and no use of tobacco or nicotine products for at least 3 months;
* Females will be non-pregnant, non-lactating, and either post-menopausal for at least 1 year, surgically sterile (including tubal ligation, hysterectomy) for at least 3 months, until 30 days following Study Completion be willing to use an approved method of contraception;
* Has normal nasal mucosa.

Exclusion Criteria:

* Previous surgical treatment for obesity;
* Serious Medical Condition
* Serious Psychiatric illness
* Organic causes of obesity (e.g. untreated hypothyroidism)
* Type 1 or Type 2 Diabetes;
* Presence of uncontrolled hypertension
* On prohibited concomitant medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of increasing nasal PYY3 36 dosing on weight loss post 24 weeks of treatment | 24 Weeks

SECONDARY OUTCOMES:
To evaluate the safety of three nasal PYY3 36 dose groups compared to nasal placebo | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Brandt, M.D., Study Director — Nastech Pharmaceutical Company, Inc.
Locations (28):
- United States (28):
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Peoria, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Anaheim, California
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Beverly Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Carmichael, California
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Sacramento, California
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, San Francisco, California
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Pembroke Pines, Florida
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Valparaiso, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Baton Rouge, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Brooklyn Center, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Manlius, New York
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Reading, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Greer, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Mt. Pleasant, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Temple, Texas
  - For additional information regarding investigative sites for this trial, contact 1-425-415-3011, Salt Lake City, Utah